CLINICAL TRIAL: NCT04181385
Title: Assessment of Lipid Response to Acute Olanzapine in Healthy Adults
Brief Title: Acute Olanzapine and Lipid Response
Acronym: OLA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: OLA 15-8951
Record Dates: First submitted 2019-11-25; First posted 2019-11-29 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: olanzapine

STUDY DESIGN:
Intervention Model Description: Participants receive either placebo, olanzapine or olanzapine plus bromocriptine, in random order on 3 separate study visits, with blood samples taken before and after treatment and intake of a high-fat drink
Who Masked: Participant
Masking Description: Single-blinded study with participant blinded to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Olanzapine (Experimental): Olanzapine, 10mg, oral, single dose
  Interventions: Drug: Olanzapine 10 milligram
- Olanzapine plus bromocriptine (Experimental): Olanzapine, 10mg, oral, single dose Bromocriptine, 5mg, oral, single dose
  Interventions: Drug: Olanzapine 10 milligram; Drug: Bromocriptine 5 milligram
- Placebo (Placebo Comparator): Placebo, oral, single dose
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Olanzapine 10 milligram — Oral olanzapine capsule
  Arms: Olanzapine; Olanzapine plus bromocriptine
Drug: Bromocriptine 5 milligram — Oral bromocriptine capsule
  Arms: Olanzapine plus bromocriptine
Drug: Placebo oral tablet — oral placebo capsules
  Arms: Placebo

SUMMARY:
Atypical antipsychotics are pharmaceutical drugs used to treat schizophrenia. Common side effects are weight gain, insulin resistance, and abnormal blood lipids. This increases the risk for type 2 diabetes and cardiovascular disease in patients taking these drugs. In particular, olanzapine is a highly effective therapy for schizophrenia but is commonly associated with metabolic disturbances. It has previously been shown that the negative effects on insulin sensitivity and glucose metabolism occur even after a single dose, independently of weight gain. These effects may be mediated by blocking the dopamine (D2) receptor. In this study the research team is investigating whether a single dose of olanzapine alters postprandial lipid metabolism after a high-fat drink. Olanzapine administered along with the high-fat drink will be compared to placebo or olanzapine plus bromocriptine (an activator of the D2 receptor).

DETAILED DESCRIPTION:
Postprandial lipid and hormonal responses are being investigated in up to 15 individuals. Participants are their own control in a single-blind, placebo-controlled, crossover design. Participants are admitted after an overnight fast. Participants will consume a high-fat drink (50g of fat) along with either oral placebo, olanzapine (10mg) or olanzapine (10mg) plus bromocriptine (5mg). Study visits occur 2-4 weeks apart with the three treatments applied in random order. Blood samples will be taken at baseline and regular intervals after the treatments for up to 8 hours to measure glucose, insulin, triglycerides, fatty acids and other hormones/metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 60 years
* Body mass index (BMI) 20 to 40 kg/m2
* Hemoglobin in the normal range.
* Normal glucose tolerance in response to a 75 gram, 2-hr oral glucose tolerance test
* Women of reproductive age should be on contraception (oral contraceptive pill or intra-uterine device/coil) for at least 2 months prior to and after the study. Anyone with a positive urine pregnancy test (carried out at screening and the day before each kinetic study) will be excluded.

Exclusion Criteria:

* Any volunteer with evidence of prolonged corrected QT interval (>470 ms in males and >450ms in females)
* Any volunteer with morbid obesity (BMI>40 or BMI>30 with any obesity related medical complication such as diabetes, hypertension or coronary disease)
* Any history of a myocardial infarction or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on echocardiogram, unstable angina, or decompensated heart failure
* Study participant with a history of hepatic disease that has been active within the previous two years.
* Any current or previous history of biliary disease (including gall stones, biliary atresia and cholecystitis) or pancreatitis.
* Any current or previous history of endocrine disease, dyslipidemia or malignancy
* Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL) genitourinary, hematological systems, or has severe uncontrolled treated or untreated hyper/ hypotension (sitting diastolic BP > 100 or systolic > 180 or systolic BP<100) or proliferative retinopathy
* Use of immunosuppressive agents at any time during the study
* Allergy to any study medication
* Pregnancy (as ascertained by urinary human chorionic gonadotropin at screening and the day before each study visit) or breastfeeding
* Fasting blood glucose > 6.0 mmol/l or known diabetes.
* Any laboratory values: aspartate aminotransferase > 2x upper limit of normal (ULN); alanine transaminase >2x ULN thyroid stimulating hormone > 6 mU/l
* Current addiction to alcohol or substances of abuse as determined by the investigator or of any mental illness.
* Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
* Taking any regular prescription or non-prescription medications at the time of the study. Occasional use of medications such as acetaminophen or Tylenol 1 or any use of natural health products may be permitted at the discretion of the investigator.
* Will not donate blood three months prior to and three months post study procedures
* Hemoglobin below the reference range (less than 130 g/l for males and 120 g/l for females) based on blood tests at screening and on the day before the kinetic study
* Hematocrit below the reference range (less than 0.38 for males and 0.37 for females) based on blood tests at screening and on the day before the kinetic study
* Soy allergy (component of high-fat drink)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Plasma triglycerides | 8 hours
  Plasma triglycerides measured after treatments
Plasma fatty acids | 8 hours
  Plasma fatty acids measured after treatments

CONTACTS AND LOCATIONS:
Overall Officials: Satya Dash, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No